CLINICAL TRIAL: NCT02213432
Title: Randomized Controlled Trial to Compare Seroprotection Rate According to Timing of Influenza Vaccination in Adult Patients With Non-Hematologic Malignancies Receiving Scheduled Cytotoxic Chemotherapy
Brief Title: Influenza Vaccination in Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Seoul National University Hospital (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Principal Investigator, Wan Beom Park, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1407-057-593
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Cancer
Keywords: influenza vaccine; cancer
MeSH Terms: conditions — Neoplasms; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day 1 vaccination (Experimental): Different timing of influenza vaccination: Day 1
  Day 1 vaccination group: patients will be vaccinated against influenza at the day (Day 1) when chemotherapy starts.
  Interventions: Biological: Different timing of influenza vaccination
- Day 11 vaccination (Active Comparator): Different timing of influenza vaccination: Day 11
  Day 11 vaccination group: patients will be vaccinated against influenza at the 11th days after chemotherapy starts
  Interventions: Biological: Different timing of influenza vaccination

INTERVENTIONS:
Biological: Different timing of influenza vaccination — The timing of Influenza vaccination for cancer patients receiving chemotherapy will be differently assigned to day 1 or day 11.

SUMMARY:
The purpose of this study is to determine the timing of influenza vaccination to induce higher antibody response in adult patients with non-hematologic malignancies receiving scheduled cytotoxic chemotherapy.

DETAILED DESCRIPTION:
The participants will be stratified by the age (cut off; 60 years old) and last year influenza vaccination, and block-randomized to 2 groups; Day 1 vaccination group and Day 11 vaccination group.

Day 1 group will be vaccinated at Day 1, when the cycle of chemotherapy begins. Day 11 group will get the vaccine at Day 11, 10 days after chemotherapy begins.

As the rate of completion of study in the Day 11 group is anticipated lower than Day 1 group, we will assign the participants into Day 1: Day 11 with the different ratio; 4:5.

Hemagglutination inhibition Ab titre at pre-vaccination and post-vaccination (21-28 days after vaccination) will be examined in all participants.

All the participants will be asked if they have any contraindication for influenza vaccine by a physician before vaccination. And they will be monitored for any adverse reaction of the vaccination after 2-4 days(phone calling) and after 21-28 days (visiting the hospital).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who receive the scheduled cytotoxic chemotherapy every 3 weeks because of solid cancer.

   Specific definition of each term is like following:
   * The solid cancer includes various kinds of cancer except hematologic and lymphoid malignancies.
   * Cytotoxic chemotherapy includes adjuvant, neoadjuvant or palliative purpose of chemotherapy with the planned duration at least over 3 cycles every 3 weeks.
   * Targeted therapy drugs like as monoclonal antibody, tyrosine kinase inhibitor or oral chemotherapy drugs like as Xeloda are excluded.
2. Patients who did not receive the influenza vaccination yet in the current year.
3. Older than 19 years
4. Eastern Cooperative Oncology Group (ECOG) performance status is 0, 1, or 2
5. Cell blood count meets following criteria:

   * Neutrophile count ≥ 1.5 x 10^9/L
   * Platelet count ≥ 100 x 10^9/L
   * Hemoglobin ≥ 8 g/dL
6. Patients who can understand and agreed with the informed consents.

Exclusion Criteria:

1. Patients who have any contraindication for influenza vaccination.
2. Patients who are supposed to receive the last chemotherapy at the enrollment
3. Patients who receive simultaneous radiation therapy with cytotoxic chemotherapy
4. Patients who receive any immunosuppressant (excluding steroid for anti-emetic effect)
5. Patients with HIV and low CD 4+ T cell count (< 500/uL)
6. Patients with autoimmune disease who are anticipated to have a problem with immunogenicity for vaccine
7. Patients who have transplanted organ and receive immunosuppressants
8. Patients who are supposed to get prophylactic G-CSF after chemotherapy
9. Patients who are suspected to have active infectious disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate | 21-28 days after vaccination
  The percentage of vaccine recipients with a serum haemagglutination inhibition(HI) titre ≥40 post vaccination (21-28 days)

SECONDARY OUTCOMES:
Seroconversion factor | 21-28 days after vaccination
  Seroconversion factor is defined as mean fold increases in geometric mean titers of the haemagglutination inhibition(HI) after vaccination, expressed as a multiple.
Seroconversion rate | 21-28 days after vaccination
  Seroconversion rate is defined as the percentage of vaccine recipients with a fourfold increase or more in post-vaccination HI titre
Geometric mean titre of HI | 21-28 days after vaccination
  Geometric mean titers of HI (haemagglutination inhibition) after vaccination
Vaccine-related adverse events | within 28 days
  the proportion of patients with any or serious vaccine-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wan Beom Park, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea